| Da | idy ID<br>te<br>ne | |
|---|---|---|
| | CONSENT FORM | |
| Titl | e of Project: Resilience Training for Surgeons | |
| Na | me of Researcher: Mr Stephen Richer | |
| | Please initi | al all boxes |
| 1. | I confirm that I have read and understand the information sheet dated 15/01/18(version 1.1) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from the research team, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |
| 4. | I understand that my name will not be linked with the research materials, and I will not be identified or identifiable in the outputs that result from the research. | |

IRAS: 238751 15/01/18 Version 1.2 IRAS: 238751 15/01/18 Version 1.2

| 5. | I understand taking part<br>that these recordings wi<br>independent ACT asses | t by an appropriate | |
|---|---|---|---|
| 6. | I agree to take part in the | e above study. | |
| —<br>Nai | me of Participant | <br>Date | Signature |
| | me of Person<br>ng consent. | <br>Date | Signature |

This form should be signed and dated by all parties after the participant receives a copy of the participant information sheet and any other written information provided to the participants. A copy of the signed and dated participant agreement form should be kept with the project's main documents which must be kept in a secure location.